CLINICAL TRIAL: NCT05195528
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Vonoprazan 10 and 20 mg Compared to Placebo for Relief of Heartburn in Subjects With Symptomatic Non-Erosive Gastroesophageal Reflux Disease (NERD) After 4 Weeks and to Evaluate the Efficacy and Safety of Vonoprazan 10 and 20 mg for Relief of Heartburn in Subjects With NERD After 6 Months
Brief Title: A Study to Evaluate the Efficacy and Safety of Vonoprazan Compared to Placebo for Relief of Heartburn in Participants With Symptomatic Non-Erosive Gastroesophageal Reflux Disease (NERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NERD-301
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Non-Erosive Gastro-Esophageal Reflux Disease; Heartburn
Keywords: NERD; Vonoprazan
MeSH Terms: conditions — Heartburn | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vonoprazan 10 mg (Experimental): Participants will be administered vonoprazan at a dose of 10 mg QD in the 4 week Placebo-controlled Treatment Period. Participants randomized to vonoprazan 10 mg in the Placebo-controlled Treatment Period will continue to take the same dose in the 20 week Extension Period.
  Interventions: Drug: Vonoprazan
- Vonoprazan 20 mg (Experimental): Participants will be administered vonoprazan at a dose of 20 mg QD in the 4 week Placebo-controlled Treatment Period. Participants randomized to vonoprazan 20 mg in the Placebo-controlled Treatment Period will continue to take the same dose in the 20 week Extension Period.
  Interventions: Drug: Vonoprazan
- Placebo (Placebo Comparator): Participants will be administered the placebo QD in the 4 week Placebo-controlled Treatment Period. Participants randomized to placebo in the Placebo-controlled Treatment Period will be re-randomized to receive either vonoprazan 10 mg QD or vonoprazan 20 mg QD in the 20 week Extension Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vonoprazan — Orally via capsule
  Arms: Vonoprazan 10 mg; Vonoprazan 20 mg
Drug: Placebo — Orally via capsule
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to assess the efficacy of vonoprazan (10 mg and 20 mg once daily [QD]) compared to placebo (QD) in relief of heartburn over 4 weeks in participants with NERD.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is ≥18 years of age at the time of informed consent signing.
2. In the opinion of the investigator or subinvestigators, the participant is capable of understanding and complying with protocol requirements, including compliance with the electronic diary.
3. The participant signs and dates a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures. The participant is informed of the full nature and purpose of the study, including possible risks and side effects. The participant has the ability to cooperate with the investigator. Ample time and opportunity should be given to read and understand verbal and/or written instructions.
4. The subject has a diagnosis of symptomatic gastroesophageal reflux disease (GERD) with heartburn as the subject's predominant symptom prior to the Screening Period, as documented in the subject's medical record.
5. History of onset of heartburn at least 6 months prior to the Screening Period.
6. Heartburn reported on 4 or more days during any consecutive 7-day period of the Screening Period as recorded in the electronic diary.
7. A female participant of childbearing potential who is or may be sexually active with a non-sterilized male partner agrees to routinely use adequate contraception from the signing of informed consent until 4 weeks after the last dose of study drug.

Exclusion Criteria:

1. The participant has endoscopically confirmed erosive esophagitis (EE) during the Screening Period. Endoscopy conducted during the Screening Period should be performed after participants meet Inclusion Criterion 6 (i.e., heartburn reported on 4 or more days during any consecutive 7-day period of the Screening Period as recorded in the electronic diary).
2. The participant has active irritable bowel syndrome (IBS) or has had a flare of IBS requiring therapy within the prior 6 months.
3. The participant has a history of or is suspected of having functional upper gastrointestinal disorders, such as:

   1. Functional heartburn, as described in the Rome IV Criteria.
   2. Functional dyspepsia, as described in the Rome IV Criteria.
4. The participant has endoscopic Barrett's esophagus (>1 cm of columnar-lined esophagus) and/or definite dysplastic changes in the esophagus.
5. The participant has any other clinically significant condition affecting the esophagus, including eosinophilic esophagitis; esophageal varices; viral or fungal infection; esophageal stricture; a history of radiation therapy, radiofrequency ablation, endoscopic mucosal resection, or cryotherapy to the esophagus; or any history of caustic or physiochemical trauma (including sclerotherapy or esophageal variceal band ligation). However, participants diagnosed with Schatzki's ring (mucosal tissue ring around lower esophageal sphincter) or hiatal hernia are eligible to participate.
6. The participant has scleroderma (systemic sclerosis) or systemic lupus erythematosus.
7. The participant has a history of surgery or endoscopic treatment affecting gastroesophageal reflux, including fundoplication and dilation for esophageal stricture (except dilation for a Schatzki's ring) or a history of gastric or duodenal surgery (except endoscopic removal of benign polyps).
8. The participant has an active gastric or duodenal ulcer within 4 weeks before the first dose of study drug.
9. The participant requires or is expected to require use of prescription or non-prescription proton pump inhibitors (PPIs) or histamine-2 receptor antagonists (H2RAs) throughout the study.
10. The participant has received any investigational compound (including those in post-marketing studies) within 30 days prior to the start of the Screening Period or vonoprazan in a clinical trial at any time (including participation in Study NERD-201). A participant who has been screen failed from another clinical study and who has not been dosed may be considered for enrollment in this study.
11. The participant is a study site employee, an immediate family member, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or who may have consented under duress.
12. The participant has had clinically significant upper or lower gastrointestinal bleeding within 4 weeks prior to the Screening Period.
13. The participant has Zollinger-Ellison syndrome or other gastric acid hypersecretory conditions.
14. The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, and titanium oxide, or red or yellow ferric oxide). Skin testing may be performed according to local standard practice to confirm hypersensitivity.
15. The participant has a history of alcohol abuse, illegal drug use, or drug addiction within the 12 months prior to screening, or regularly consumes >21 units of alcohol (1 unit = 12 oz/300 mL beer, 1.5 oz/25 mL hard liquor/spirits, or 5 oz/100 mL wine) per week based on self-report. Participants must have a negative urine drug screen for cannabinoids/tetrahydrocannabinol (including prescription cannabinoids) and non-prescribed medications during the Screening Period.
16. The participant is taking any excluded medications or treatments listed in the protocol, including prescription cannabinoids/tetrahydrocannabinol.
17. If female, the participant is pregnant, lactating, or intending to become pregnant before, during, or within 4 weeks after participating in this study, or intending to donate ova during such time period.
18. The participant has a history or clinical manifestations of significant central nervous system, cardiovascular, pulmonary, hepatic, renal, metabolic, other gastrointestinal, urological, endocrine, or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participant safety.
19. The participant requires hospitalization or has surgery scheduled during the course of the study (from Visit 1 to end of Follow-up Period at Visit 10) or has undergone major surgical procedures within 30 days prior to the Screening Period.
20. The participant has a history of malignancy (including mucosa-associated lymphoid tissue lymphoma) or has been treated for malignancy within 5 years prior to the start of the Screening Period (Visit 1). (The participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
21. The participant has acquired immunodeficiency syndrome or human immunodeficiency virus infection, or tests positive for the hepatitis B surface antigen, hepatitis C virus (HCV) antibody, or HCV-ribonucleic acid (RNA). However, participants who test positive for HCV antibody but negative for HCV-RNA are permitted to participate.
22. The participant has any of the following abnormal laboratory test values at the start of the Screening Period:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >2 × ULN (except for participants with a diagnosis of Gilbert's syndrome).
23. The subject tests positive for active H pylori infection during the Screening Period, after ≥4 weeks free from antibiotics and bismuth and ≥2 weeks free from PPIs and histamine-2 receptor antagonists (H2RAs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (108):
- United States (108):
  - North Alabama Research Center LLC, Athens, Alabama
  - Cullman Research Center, Cullman, Alabama
  - Medical Affiliated Research Center Inc, Huntsville, Alabama
  - East View Medical Research, LLC, Mobile, Alabama
  - Elite Clinical Studies - Phoenix - Clinedge, Phoenix, Arizona
  - Del Sol Research Management - Clinedge, Tucson, Arizona
  - Preferred Research Partners - ClinEdge, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Alliance Research Institute, Canoga Park, California
  - GW Research, Inc, Chula Vista, California
  - eStudy Site, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - BG Clinical Research, Encinitas, California
  - Paragon Rx Clinical, Garden Grove, California
  - OM Research LLC, Lancaster, California
  - Torrance Clinical Research Institute, Lomita, California
  - Prospective Research Innovations, Rancho Cucamonga, California
  - Northern California Research Corp, Sacramento, California
  - Digestive Care Center, San Carlos, California
  - Clinical Applications Laboratories Inc, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Paragon Rx Clinical, Inc., Santa Ana, California
  - Western States Clinical Research Inc, Wheat Ridge, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Velocity Clinical Research - New Smyrna Beach, Edgewater, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - ENCORE Borland-Groover Clinical Research, Jacksonville, Florida
  - ClinCloud, Maitland, Florida
  - Legacy Clinical Solutions: Sensible HealthCare, LLC, Ocoee, Florida
  - Digestive Disease Consultants, PA, Orange Park, Florida
  - Medical Center, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Guardian Angel Research, Tampa, Florida
  - Southeast Clinical Research Center, Dalton, Georgia
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Atlanta Center For Clinical Research, Roswell, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - In Quest Medical Research, Suwanee, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Iowa Digestive Disease Center, Clive, Iowa
  - Kansas Medical Clinic, Topeka, Kansas
  - Clinical Trials Management LLC, Covington, Louisiana
  - Combined Gastro Research, Lafayette, Louisiana
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Clinical Trials of America, LLC, West Monroe, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Digestive Health Specialists, Chelmsford, Massachusetts
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - MNGI Digestive Health, Minneapolis, Minnesota
  - Minnesota Gastroenterology PA, Plymouth, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Quality Clinical Research - HyperCore, Omaha, Nebraska
  - Sierra Clinical Research, Las Vegas, Nevada
  - Office of Site 1, Las Vegas, Nevada
  - Office of Site 2, Las Vegas, Nevada
  - Advanced Research Institute, Reno, Nevada
  - The Gastroenterology Group of Northern NJ LLC, Englewood, New Jersey
  - Allied Health Clinical Research Organization, Freehold, New Jersey
  - NY Scientific, Brooklyn, New York
  - Drug Trials America, Hartsdale, New York
  - Care Access Research, New York, New York
  - UNC Medical Center, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology PLLC, Charlotte, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Clinical Trials of America-NC, LLC, Mount Airy, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Gastro Health Research, Cincinnati, Ohio
  - Remington Davis Clinical Research, Columbus, Ohio
  - Great Lakes Medical Research LLC, Mentor, Ohio
  - North Shore Gastroenterology, Westlake, Ohio
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Gastroenterology Associates, PA of Greenville, Greenville, South Carolina
  - Gastro One, Cordova, Tennessee
  - Galen Medical Group, Hixson, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - QUALITY Medical Research, Nashville, Tennessee
  - Vanderbilt Digestive Disease Center, Nashville, Tennessee
  - Gastroenterology Consultants of South Texas, PLLC, Brownsville, Texas
  - Digestive Health Associates of Texas, PA, Carrollton, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - Texas Tech Physicians of El Paso, El Paso, Texas
  - Digestive Health Associates of Texas, P.A.dba DHAT Research Institute, Garland, Texas
  - Primecare Medical Group, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Quality Research Inc, San Antonio, Texas
  - Gastroenterology Research of San Antonio (GERSA), San Antonio, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - GI Alliance, Southlake, Texas
  - Texas Gastro Consultants, Tomball, Texas
  - Advanced Research Institute, Ogden, Utah
  - Kalo Clinical Research, Salt Lake City, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Clinical Research Partners LLC, Richmond, Virginia
  - Washington Gastroenterology, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antunes C, Ghosh G, Katz P, Yadlapati R, Leifke E, Harris T, Graham H, Laine L. Vonoprazan Improves Nocturnal Gastroesophageal Reflux Symptoms in Nonerosive Reflux Disease. Am J Gastroenterol. 2025 Oct 13. doi: 10.14309/ajg.0000000000003794. Online ahead of print. PMID 41081570
- [Derived] Laine L, Spechler S, Yadlapati R, Schnoll-Sussman F, Smith N, Leifke E, Harris T, Hunt B, Fass R, Katz P. Vonoprazan is Efficacious for Treatment of Heartburn in Non-erosive Reflux Disease: A Randomized Trial. Clin Gastroenterol Hepatol. 2024 Nov;22(11):2211-2220.e10. doi: 10.1016/j.cgh.2024.05.004. Epub 2024 May 14. PMID 38750866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 91 sites in the United States in the period of time from January 2022 to May 2023. Participants were in the study for a period of time up to 33 weeks.
Pre-assignment Details: Participant were randomized in a 1:1:1 ratio to receive vonoprazan 10 mg , vonoprazan 20 mg, or placebo during the Part 1 Placebo-controlled Treatment Period. In the Part 2 Extension Period participants who had been assigned vonoprazan in Part 1 continued with their assigned treatment while those assigned placebo in Part 1 were re-randomized to receive vonoprazan 10 mg or 20 mg.
Groups:
- Placebo: Participants with Non-Erosive Gastroesophageal Reflux Disease (NERD) and heartburn symptoms were randomized to receive placebo once per day (QD) for 4 weeks during the Part 1 Placebo-controlled Treatment Period.
- Vonoprazan 10 mg: Participants with NERD and heartburn symptoms were randomized to receive vonoprazan 10 mg QD for 4 weeks during the Part 1 Placebo-controlled Treatment Period. Participants could continue taking vonoprazan 10 mg for an additional 20 weeks in the Part 2 Extension Period.
- Vonoprazan 20 mg: Participants with NERD and heartburn symptoms were randomized to receive vonoprazan 20 mg QD for 4 weeks during the Part 1 Placebo-controlled Treatment Period. Participants continued taking vonoprazan 20 mg for an additional 20 weeks in the Part 2 Extension Period.
- Placebo/Vonoprazan 10 mg: Participants randomized to placebo during the Part 1 Placebo-controlled Treatment Period were re-randomized to receive vonoprazan 10 mg for 20 weeks in the Part 2 Extension Period.
- Placebo/Vonoprazan 20 mg: Participants randomized to placebo during the Part 1 Placebo-controlled Treatment Period were re-randomized to receive vonoprazan 20 mg for 20 weeks in the Part 2 Extension Period.
Period: Placebo-controlled Treatment Period
Arm/Group | Placebo | Vonoprazan 10 mg | Vonoprazan 20 mg | Placebo/Vonoprazan 10 mg | Placebo/Vonoprazan 20 mg
Started | 259 | 258 | 259 | 0 | 0
Intent to Treat Analysis Set (Intent-to-treat (ITT): all efficacy analyses were conducted on the ITT Set using the planned treatment even if the participant received a different incorrect treatment.) | 258 | 257 | 257 | 0 | 0
Safety Analysis Set (Safety Analysis Set (SAS): all safety analyses were conducted on the Safety Set using the actual treatment the participant received even if the participant was randomized to receive a different treatment.) | 256 | 259 (Planned and actual treatment differed for 2 participants.) | 257 | 0 | 0
Completed | 247 | 250 | 242 | 0 | 0
Not Completed | 12 | 8 | 17 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — Pre-Treatment Event (PTE) or Adverse Event (AE) or Serious Adverse Event (SAE) | 2 | 1 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 4 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Not Treated | 1 | 1 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: Extension Period
Arm/Group | Placebo | Vonoprazan 10 mg | Vonoprazan 20 mg | Placebo/Vonoprazan 10 mg | Placebo/Vonoprazan 20 mg
Started | 0 | 247 | 237 | 122 | 122
Intent to Treat Analysis Set (ITT: all efficacy analyses were conducted on the ITT Set using the planned treatment even if the participant received a different incorrect treatment.) | 0 | 247 | 235 | 119 | 122
Safety Analysis Set (SAS: all safety analyses were conducted on the Safety Set using the actual treatment the participant received even if the participant was randomized to receive a different treatment.) | 0 | 248 (Planned and actual treatment differed for 1 participant.) | 236 (Planned and actual treatment differed for 1 participant.) | 118 | 121
Completed | 0 | 219 | 206 | 106 | 103
Not Completed | 0 | 28 | 31 | 16 | 19
Not completed — PTE or AE or SAE | 0 | 4 | 5 | 4 | 4
Not completed — Protocol Violation | 0 | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 6 | 13 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 12 | 9 | 6 | 5
Not completed — Lack of Efficacy | 0 | 3 | 0 | 0 | 2
Not completed — Not Treated | 0 | 0 | 2 | 3 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data is presented for the Placebo-controlled treatment Period, ITT population.
Groups:
- Placebo: Participants with NERD and heartburn symptoms were randomized to receive placebo QD for 4 weeks during the Part 1 Placebo-controlled Treatment Period.
- Vonoprazan 10 mg: Participants with NERD and heartburn symptoms were randomized to receive vonoprazan 10 mg QD for 4 weeks during the Part 1 Placebo-controlled Treatment Period.
- Vonoprazan 20 mg: Participants with NERD and heartburn symptoms were randomized to receive vonoprazan 20 mg QD for 4 weeks during the Part 1 Placebo-controlled Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Vonoprazan 10 mg | Vonoprazan 20 mg | Total
Number analyzed (Participants) | 258 | 257 | 257 | 772
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (14.74) | 51 (14.03) | 50.4 (14.39) | 50.9 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 182 | 166 | 527
  Male | 79 | 75 | 91 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 87 | 80 | 244
  Not Hispanic or Latino | 180 | 165 | 171 | 516
  Unknown or Not Reported | 1 | 5 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 12 | 22 | 11 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 33 | 38 | 52 | 123
  White | 205 | 186 | 185 | 576
  More than one race | 3 | 4 | 4 | 11
  Unknown or Not Reported | 4 | 4 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Without Daytime or Nighttime Heartburn
Description: Participants were assigned an electronic diary to complete twice daily, in the morning and evening. Diary day was considered heartburn-free if both morning and evening diary entries were heartburn-free and there was no reported use of rescue antacid, H2RAs, or PPIs.
Time Frame: Day 1 to Day 28
Population: Intent-to-treat (ITT) was defined as all participants randomized into the placebo-controlled treatment period who received at least one dose of study drug and had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Placebo | Vonoprazan 10 mg | Vonoprazan 20 mg
Number analyzed (Participants) | 256 | 256 | 257
Percentage of days | 27.7 [23.92 to 31.46] | 44.8 [41.06 to 48.58] | 44.4 [40.62 to 48.15]
Statistical Analysis 1: Comparison: Placebo vs Vonoprazan 10 mg; Test type: Superiority; p < 0.0001, General linear model — P-values were obtained from the general linear model with treatment group as factor and severity and frequency of heartburn at baseline as covariates; Difference in least square mean = 17.1, 95% CI 2-sided [11.81 to 22.45]
Statistical Analysis 2: Comparison: Placebo vs Vonoprazan 20 mg; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = 16.7, 95% CI 2-sided [11.36 to 22.04]

2. Secondary Outcome: Percentage of Days Without Rescue Antacid Use
Description: Participants were assigned an electronic diary to complete twice daily, in the morning and evening. Participants recorded use of rescue antacid.
Time Frame: Day 1 to Day 28
Population: ITT was defined as all participants randomized into the placebo-controlled treatment period who received at least one dose of study drug and had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Placebo | Vonoprazan 10 mg | Vonoprazan 20 mg
Number analyzed (Participants) | 256 | 254 | 257
Percentage of days | 47.6 [43.43 to 51.68] | 63.3 [59.19 to 67.45] | 61.2 [57.12 to 65.36]
Statistical Analysis 1: Comparison: Placebo vs Vonoprazan 10 mg; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = 15.8, 95% CI 2-sided [9.93 to 21.60]
Statistical Analysis 2: Comparison: Placebo vs Vonoprazan 20 mg; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = 13.7, 95% CI 2-sided [7.84 to 19.54]

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from time of enrollment through 33 weeks (5 weeks screening, 4 weeks Placebo-controlled Treatment Period, 20 weeks Extension Period, 4 weeks follow-up). Treatment-emergent adverse events were collected from first dose of study treatment through 28 weeks.
Description: All-cause mortality was summarized for all enrolled participants. Serious and Other Adverse Events were summarized in the SAS, which includes randomized subjects who received at least one dose of study drug.
Groups:
- Placebo (Part 1: 4 Weeks): Participants with NERD and heartburn symptoms were randomized to receive placebo QD for 4 weeks during the Part 1 Placebo-controlled Treatment Period.
- Vonoprazan 10 mg (Part 1: 4 Weeks): Participants with NERD and heartburn symptoms were randomized to receive vonoprazan 10 mg QD for 4 weeks during the Part 1 Placebo-controlled Treament Period.
- Vonoprazan 20 mg (Part 1: 4 Weeks) Part 1: Participants with NERD and heartburn symptoms were randomized to receive vonoprazan 20 mg QD for 4 weeks during the Part 1 Placebo-controlled Treament Period.
- Placebo/Vonoprazan 10 mg (Part 2: 20 Weeks); Vonoprazan 10 mg/Vonoprazan 10 mg (Part 2: 20 Weeks): Participants randomized to placebo during the Part 1 Placebo-controlled Treatment Period were re-randomized to receive vonoprazan 10 mg for 20 weeks in the Part 2 Extension Period.
- Placebo/Vonoprazan 20 mg (Part 2: 20 Weeks); Vonoprazan 20/Vonoprazan 20 mg (Part 2: 20 Weeks): Participants randomized to placebo during the Part 1 Placebo-controlled Treatment Period were re-randomized to receive vonoprazan 20 mg for 20 weeks in the Part 2 Extension Period.
Arm/Group | Placebo (Part 1: 4 Weeks) | Vonoprazan 10 mg (Part 1: 4 Weeks) | Vonoprazan 20 mg (Part 1: 4 Weeks) Part 1 | Placebo/Vonoprazan 10 mg (Part 2: 20 Weeks) | Placebo/Vonoprazan 20 mg (Part 2: 20 Weeks) | Vonoprazan 10 mg/Vonoprazan 10 mg (Part 2: 20 Weeks) | Vonoprazan 20/Vonoprazan 20 mg (Part 2: 20 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/258 | 0/259 | 0/122 | 0/122 | 0/247 | 0/237
Serious Adverse Events (participants affected / at risk) | 0/256 | 1/259 | 2/257 | 2/118 | 4/121 | 7/248 | 3/236
Other Adverse Events (participants affected / at risk) | 17/256 | 28/259 | 32/257 | 26/118 | 11/121 | 40/248 | 45/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part 1: 4 Weeks) (N=256) | Vonoprazan 10 mg (Part 1: 4 Weeks) (N=259) | Vonoprazan 20 mg (Part 1: 4 Weeks) Part 1 (N=257) | Placebo/Vonoprazan 10 mg (Part 2: 20 Weeks) (N=118) | Placebo/Vonoprazan 20 mg (Part 2: 20 Weeks) (N=121) | Vonoprazan 10 mg/Vonoprazan 10 mg (Part 2: 20 Weeks) (N=248) | Vonoprazan 20/Vonoprazan 20 mg (Part 2: 20 Weeks) (N=236)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part 1: 4 Weeks) (N=256) | Vonoprazan 10 mg (Part 1: 4 Weeks) (N=259) | Vonoprazan 20 mg (Part 1: 4 Weeks) Part 1 (N=257) | Placebo/Vonoprazan 10 mg (Part 2: 20 Weeks) (N=118) | Placebo/Vonoprazan 20 mg (Part 2: 20 Weeks) (N=121) | Vonoprazan 10 mg/Vonoprazan 10 mg (Part 2: 20 Weeks) (N=248) | Vonoprazan 20/Vonoprazan 20 mg (Part 2: 20 Weeks) (N=236)
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 6 | 2 | 1 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 6 | 2 | 1 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 1 | 2 | 2 | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 6 | 8 | 1 | 1 | 3 | 5
COVID-19 (Infections and infestations) | 2 | 3 | 4 | 12 | 3 | 11 | 20
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 1 | 5 (5)
Influenza (Infections and infestations) | 1 | 0 | 1 | 4 | 2 | 5 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1 | 5 | 2 | 0 | 0 | 5
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 2 | 2 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 1 | 12 | 5
Urinary tract infection (Infections and infestations) | 3 | 4 | 4 | 2 | 0 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT05195528/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT05195528/SAP_001.pdf